CLINICAL TRIAL: NCT02071875
Title: A Non-Randomized, Non-Significant Risk Study Comparing the Nautilus NeuroWaveTM System to Transcranial Doppler or DSA as an Aid to Diagnosing Vasospasm
Brief Title: Comparing the Nautilus NeuroWaveTM to TCD or DSA for the Detection of Vasospasm
Status: Terminated | Type: Observational
Why Stopped: Study recruitment was put on hold for interim data analysis and during this time period the PI requested to pre-maturely terminate the study
Sponsor: Jan Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NMDCL100212-OCA
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Vasospasm
Keywords: Vasospasm; Aneurysm; SAH; Nautilus NeuroWave
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nautilus NeuroWaveTM recording: Nautilus NeuroWaveTM recording 15 minute recording
  Interventions: Device: Nautilus NeuroWaveTM recording

INTERVENTIONS:
Device: Nautilus NeuroWaveTM recording — Nautilus NeuroWaveTM recording 15 minute recording with Nautilus NeuroWave Neurodiagnostic .

SUMMARY:
To determine the efficacy of using the Jan Medical NNW system as a diagnostic aid in detection of moderate and severe vasospasm for detection of vasospasm in patients with subarachnoid hemorrhage.

DETAILED DESCRIPTION:
This study is a prospective, comparative, non-randomized study in subjects with subarachnoid hemorrhage who are undergoing surveillance for vasospasm. The study will be conducted in one center.

The primary objective of Phase I of this non-significant risk study is proof of principle. During this phase the goal is to build a library of Jan Medical NNW system recordings from patients with moderate and severe vasospasms. A signature for detecting vasospasms will be developed using the signals from a vasospasm epoch to a patient's individual baseline recording and confirming the presence of vasospasm by comparison of Jan Medical NNW system data to TCD and, when available Digital Subtraction Angiography (DSA). The number of patients required for Phase I is estimated to be 20 patients with confirmed moderate or severe vasospasm with a minimum of 10 these patients having at least one severe vasospasm recording confirmed by TCD or DSA. Daily recordings are to be taken.

During Phase II the Jan Medical NNW system will independently utilize the signatures identified in Phase I to identify the presence or absence of moderate and severe vasospasm in a blinded recording. This recording will be compared to TCD or DSA, when DSA is available, for analysis of sensitivity and specificity. Up to 50 subjects will be enrolled in Phase II. When possible, multiple recordings will be obtained from each subject to include recordings with and without vasospasm.

Duration of each subject's enrollment in this study is limited to the period of time when Jan Medical NNW system recordings are performed. No additional tests or procedures will be performed during participation in this study and all other data collected (including TCD or DSA) will be based on available evaluations conducted as part of the patient's standard of care. Upon completing the last Jan Medical NNW system recording or when no further data collection is expected, the subject will be exited from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years of age or older.
2. Subjects with subarachnoid hemorrhage who are receiving clinical and diagnostic surveillance for vasospasm.
3. Signed informed consent from the patient or the patient's Legally Authorized Representative

Exclusion Criteria:

1. Unstable medical illness such that recordings might interfere with medical care.
2. Presence of head bandages or brain monitors that might physically interfere with the NNW recording device.
3. Current hemicraniectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with subarachnoid hemorrhage who are undergoing surveillance for vasospasm
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity (moderate or severe) | Within 5 minutes from end of recording
  Efficacy at identifying moderate or severe vasospasm. Reference diagnosis will be with TCD and where available DSA
Specificity | Within 5 minutes of recording
  Rate of false positives using TCD and where available DSA as the reference standard. False positive is a recording judged mild or no vasospasm by TCD or DSA that is determined by the NNW as moderate or severe

SECONDARY OUTCOMES:
Sensitivity at detecting any vasospasm | Within 5 minutes of recording
  Efficacy at identifying vasospasm either mild, moderate or severe. Reference standard will be TCD and DSA where available.
Specificity | Within 5 minutes of end of recording
  Rate of false positives using TCD and where available DSA as the reference standard. False positive is a recording determined as no vasospasm by TCD or DSA that is determined by the NNW as either mild, moderate or severe vasospasm
Location of vasospasm | Within 5 minutes of recording
  With TCD and DSA, when available, as reference standards, the efficacy at locating any vasospasm as ocurring in the left, right or back of the cranium. The measure will be what % of correctly called vasospasm was correctly located.

OTHER OUTCOMES:
Incidence of device related adverse events | Within 1 week of end of recording
  The total number of adverse events reported by the clinical site
Ease of use | Within 5 minutes from end of recording
  Number of recordings that were not of adequate quality for a determination. This will be a no call

CONTACTS AND LOCATIONS:
Overall Officials: Axel Neulen, MD, Principal Investigator — University Medical Center of the Johannes Gutenberg University Mainz
Locations (1):
- University Medical Center of the Johannes Gutenberg University Mainz, Mainz, Rhineland-Palatinate, Germany